CLINICAL TRIAL: NCT01175564
Title: A Phase I, Single Centre, Randomised, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of a Single Dose and Multiple Doses of TC-5214 (S-Mecamylamine) in Healthy Male Japanese Subjects
Brief Title: To Investigate Safety, Tolerability and Pharmacokinetics of TC-5214 in Healthy Male Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4131C00002
Record Dates: First submitted 2010-07-23; First posted 2010-08-05 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: TC-5214; safety; pharmacokinetics; single dose; repeated dose; Japanese; healthy subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Each cohort will have 9 volunteers that will receive TC-5214
  Interventions: Drug: TC-5214
- Placebo (Placebo Comparator): Each cohort will have 3 volunteers that will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5214 — Four increasing doses levels of a single dose and two increasing dose levels of 6 days repeated dose of TC-5214 tablet
  Arms: Active
Drug: Placebo — Placebo tablet, single dose and 6 days repeated dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess safety, tolerability and pharmacokinetics after a single and repeated oral doses of TC-5214 (S-mecamylamine) in healthy male Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese Healthy male ≥20 and ≤55 years old inclusive with suitable veins for cannulation or repeated venipuncture
* Have a body mass index (BMI) of ≥18 and ≤27 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* History of any clinically significant medical or neurologic disease or disorder which, in the opinion of the investigator and sponsor, may either put the subject at risk because of participation in the study, or influence the results of the subject's
* History of psychiatric disorders
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety by assessment of adverse events, brief neurological examinations, visual acuity test, vital signs, physical examinations, laboratory parameters, and electrocardiograms (ECGs), and Columbia Suicide Severity Rating Scale (C-SSRS). | Collected prior to treatment, during treatment and 7-10 days following discharge. Volunteers will be monitored througout the study for adverse events.

SECONDARY OUTCOMES:
Under Single Dosing conditions: Cmax, tmax, λz, t½λz, AUC(0-12), AUC(0-t), AUC, AUMC, MRT, % AUC extrapolated, CL/F, Vss/F, Ae fraction, Fe, (% of dose) Renal CLR. | Blood samples are taken repeatedly for 24 hours after dosing for 24 hours on Day 1 for SAD
Under Multiple Dosing Conditions: Css, max, Cmin, Cmax (tss,max), λz, t½λz, AUCss, AUC(0-t), AUC, AUMC, MRT, % AUC extrapolated, CL/F, Vss/F, Ae, Fe % of dose,Renal CLR, Rac(Cmax), Rac(AUC), Rac(Cmin)), LI, % fluctuation, time to reach the steady state | Blood samples are taken repeatedly for 24 hours after dosing for 24 hours on Day 1 for SAD and Day 6 (last dose) for MAD.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Eriksson, Study Director — AstraZeneca R&D Sodertalje, SE-151 85 Sodertalje, Sweden

REFERENCES:
- [Derived] Xu H, Henningsson A, Alverlind S, Tummala R, Toler S, Beaver JS, Al-Huniti N. Population pharmacokinetics of TC-5214, a nicotinic channel modulator, in phase I and II clinical studies. J Clin Pharmacol. 2014 Jun;54(6):707-18. doi: 10.1002/jcph.264. Epub 2014 Jan 16. PMID 24408516